CLINICAL TRIAL: NCT03240029
Title: Life Quality of Children in Cancer Remission During School Reintegration
Acronym: QdV leucémie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2009-A01379-48
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Cancer Remission
Keywords: children; life quality; school reintegration
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children in cancer remission (Experimental): Children in cancer remission sent to ordinary schools: primary (3rd, 4th, 5th grade) and middle (6th, 7th grade) schools.
  Interventions: Other: Questionnaires
- Control children (Other): Children (not in cancer remission) sent to ordinary schools (age and sex matched): primary (3rd, 4th, 5th grade) and middle (6th, 7th grade) schools.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — SPP questionnaire (Self Perception Profile for Children), Systemic inventory of life quality for children (ISQV-E), Anxiety questionnaire (STAI-C), Depression questionnaire (CDI)

SUMMARY:
Few data about the evaluation of consequences of past life with cancer on life quality of children in school reintegration are available in literature. Nevertheless, some of these studies show that the reintegration impairs life quality of these children (school difficulties, conflictual relations with peers…). The hypothesis is that children with past life with cancer have more chances to have school integration difficulties with a consequent life quality degradation compared to healthy children.

The main objective of this project is to study the relation between the satisfaction of school reintegration of children in cancer remission and the evolution of life quality in the medium term (after getting back to school). More exactly, it is the question if the satisfaction of school reintegration influences life goals and priorities of these children.

The secondary objective is to study the role of psychological status of these children (anxiety, depressive symptoms) on satisfaction-life quality relation.

A group of children with cancer history sent to ordinary school is compared to a control group of children sent to school in the same conditions (sex and age matched). Data are collected with questionnaires some months to several years after school reintegration and same questionnaires 1 year later.

If the study hypothesis is confirmed, this study will show the necessity of a long term follow up of children in cancer remission and not only medical care, but also psychological and social care, in order to support a better school reintegration.

ELIGIBILITY:
Group of children in cancer remission:

Inclusion Criteria:

* Children of both sexes in cancer remission (leukemia, with or without transplant and solid tumors), aged 8 to 12
* Stop of treatment since at least 6 months
* Back to school since some months to several years
* Signed consent of parents

Exclusion Criteria:

* Psychic difficulties
* Specialized education

Group of control children:

Inclusion Criteria:

- Signed consent of parents

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2013-09-11 (Actual); Study Completion 2013-09-11 (Actual)

PRIMARY OUTCOMES:
Life quality of children according to satisfaction of school reintegration | baseline
  Evaluated through questionnaires
Life quality of children according to satisfaction of school reintegration | 1 year
  Evaluated through questionnaires

SECONDARY OUTCOMES:
Anxiety | baseline
  Evaluated through questionnaires
Anxiety | 1 year
  Evaluated through questionnaires
Depressive symptoms | baseline
  Evaluated through questionnaires
Depressive symptoms | 1 year
  Evaluated through questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chastagner, Pr, Principal Investigator — Pediatric Hematology/Oncology, CHRU de Nancy; Fabienne Lemétayer, Study Chair — University Paul Verlaine - Metz / Human Science and art department - Health psychology team
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No